CLINICAL TRIAL: NCT03696030
Title: A Phase 1 Cellular Immunotherapy Study of Intraventricularly Administered Autologous HER2-Targeted Chimeric Antigen Receptor (HER2-CAR) T Cells in Patients With Brain and/or Leptomeningeal Metastases From HER2 Positive Cancers
Brief Title: HER2-CAR T Cells in Treating Patients With Recurrent Brain or Leptomeningeal Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17237; NCI-2018-01270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17237 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-06-27; First posted 2018-10-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Malignant Neoplasm; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Neoplasm in the Leptomeninges; Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Meningeal Carcinomatosis; Breast Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (HER2-CAR T cells) (Experimental): Patients receive HER2-CAR T cells via intraventricular administration over 5 minutes once weekly for 3 doses in the absence of disease progression or unacceptable toxicity. If patients continue to meet all eligibility criteria, they may receive additional cycles of HER2-CAR T cells at principal investigator's discretion.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given HER2-CAR T cells via intraventricular administration
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell therapy; Chimeric Antigen Receptor T-cell Infusion

SUMMARY:
This phase I trial studies the side effects and best dose of HER2-CAR T cells in treating patients with cancer that has spread to the brain or leptomeninges and has come back (recurrent). HER2-CAR T cells delivered into the ventricles of the brain may recognize and kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and recommended phase 2 dosing (RP2D) of intraventricularly administered memory-enriched autologous HER2(EQ)BBzeta/CD19t+ T cells (HER2-chimeric antigen receptor [CAR] T cells) - either HER2(EQ)BBzeta/CD19t+ TCM in Arm 1, or HER2(EQ)BBzeta/CD19t+ TN/MEM in Arm 2 - in participants with brain and/or leptomeningeal metastases from HER2 positive cancers.

SECONDARY OBJECTIVES:

I. Assess cerebrospinal fluid (CSF) and peripheral blood for HER2-CAR T cell persistence and endogenous immune system activation.

II. Describe changes in cytokine levels in the CSF and peripheral blood. III. Describe changes in circulating tumor cells in the CSF.

IV. In study participants who complete at least the first three cycles of HER2-CAR T cell infusions:

IVa. Describe the CNS clinical benefit defined as disease response rate based on Response Assessment in Neuro-Oncology Criteria (RANO) criteria (stable disease [SD], partial response [PR], or complete response [CR] in the brain).

IVb. Describe the systemic clinical benefit based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

IVc. Estimate the median central nervous system (CNS) progression-free and overall survival rates (mPFS and mOS), (newly diagnosed versus recurrent metastases).

V. In study participants who undergo tumor resection or biopsy during or after study treatment or upon autopsy, evaluate the tumor micro-environment for:

Va. HER2-CAR T cell persistence. Vb. Immune cell subsets. Vc. Cytokine levels. Vd. HER2 antigen expression levels. VI. Use biomathematical modeling of tumor growth to evaluate benefit of treatment.

OUTLINE: This is a dose-escalation study.

Patients receive HER2-CAR T cells via intraventricular administration over 5 minutes once weekly for 3 doses in the absence of disease progression or unacceptable toxicity. If patients continue to meet all eligibility criteria, they may receive additional cycles of HER2-CAR T cells at principal investigator's discretion.

After completion of study treatment, participants are followed up at 4 weeks, 3, 6, 8, 10, and 12 months, and then for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* SCREENING: Participant has treated brain and/or leptomeningeal metastases that has not recurred OR

  * Such participants are eligible to enroll in the study and undergo leukapheresis, but they cannot start treatment with HER2-CAR T cells until there is evidence of tumor progression/recurrence
* SCREENING: Participant has recurrent brain metastases after radiation therapy OR
* SCREENING: Participant has recurrent leptomeningeal metastases after intrathecal chemotherapy OR
* SCREENING: Participant has untreated brain or leptomeningeal metastases and refuses to undergo radiation and/or intrathecal chemotherapy

  * Note: Participants with leptomeningeal metastasis (diagnosed by positive CSF cytology or characteristic findings on brain or spine magnetic resonance imaging [MRI]) may have concomitant brain metastases, but having both is not required
* SCREENING: Participant must have a Karnofsky performance status (KPS) >= 70
* SCREENING: Participant must have a life expectancy of >= 8 weeks
* SCREENING: The effects of HER2-CAR T cells on a developing fetus are unknown. For this reason, women of child-bearing potential must have negative serum pregnancy test and agree to use a reliable form of birth control prior to study entry and for at least two months following duration of study participation. Male research participants must agree to use a reliable form of birth control and not donate sperm during the study and for at least six months afterwards
* SCREENING: Participant has a histologically confirmed cancer which is HER2+, defined as 3+ by immunohistochemistry (IHC) or gene amplification by fluorescence in situ hybridization (FISH)
* SCREENING: Participant must have the ability to understand and the willingness to sign a written informed consent
* ELIGIBILITY TO PROCEED WITH LEUKAPHERESIS: At least 2 weeks must have elapsed since the participant received his/her last dose of prior targeted agents, chemotherapy or radiation; at the PI's discretion, exception can be made for investigational agents that are delivered locally into the CSF
* ELIGIBILITY TO PROCEED WITH LEUKAPHERESIS: Research participant must not require more than 6 mg/day of dexamethasone (or the equivalent dose of another corticosteroid) on the day of leukapheresis
* ELIGIBILITY TO PROCEED WITH LEUKAPHERESIS: Participant must be willing to undergo placement of a catheter for central venous access if s/he does not have adequate peripheral venous access for collection of T cells
* ELIGIBILITY TO PROCEED WITH RICKHAM RESERVOIR PLACEMENT: Creatinine < 1.6 mg/dL
* ELIGIBILITY TO PROCEED WITH RICKHAM RESERVOIR PLACEMENT: White blood cell (WBC) > 2,000/uL (or absolute neutrophil count [ANC] > 1,000)
* ELIGIBILITY TO PROCEED WITH RICKHAM RESERVOIR PLACEMENT: Platelets >= 100,000/uL
* ELIGIBILITY TO PROCEED WITH RICKHAM RESERVOIR PLACEMENT: International normalized ratio (INR) must be < 1.3
* ELIGIBILITY TO PROCEED WITH RICKHAM RESERVOIR PLACEMENT: Bilirubin < 1.5 mg/dL
* ELIGIBILITY TO PROCEED WITH RICKHAM RESERVOIR PLACEMENT: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 X upper limits of normal
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Participant must be taking =< 6 mg/ day of dexamethasone (or the equivalent dose of another corticosteroid) during CAR T cell therapy
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Participants agrees to stop treatment with chemotherapy or endocrine therapy during the first 3 cycles of the HER2-CAR T cell study
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Participant does not have evidence of active infection and does not have a fever exceeding 38.5 degrees C; there is an absence of positive blood culture for bacteria, fungus, or virus within 48-hours prior to HER2-CAR T cell infusion and/or there aren't any indications of meningitis
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: WBC > 2,000/uL (or ANC > 1,000)
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Platelets > 100,000/uL. However, if platelet level is between 75,000-99,000/uL then HER2-CAR T-cell administration may proceed after platelet transfusion is given, and the post transfusion platelet count is >= 100,000/uL
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Serum creatinine < 1.8 mg/dL
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Serum total bilirubin or transaminases does not exceed 2 X upper limits of normal
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Research participant does not require supplemental oxygen to keep saturation greater than 95% and/or does not have presence of any radiographic abnormalities on chest x-ray that are positive
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Research participant does NOT have any known history of congestive heart failure (CHF) or cardiac symptoms consistent with New York Heart Association (NYHA) classification III-IV within 6 months prior to day 1 of protocol treatment, cardiomyopathy, myocarditis, myocardial infarction (MI), exposure to cardiotoxic medications or with clinical history suggestive of the above must have an electrocardiogram (EKG) and echocardiogram (ECHO) performed within 42 days prior to registration and as clinically indicated while on treatment

  * If the research participant has new symptoms of congestive heart failure (CHF), cardiomyopathy, myocarditis, MI, or exposure to cardiotoxic medications, they already had a cardiac consultation, creatinine phosphokinase (CPK), and troponin testing at pre study deeming them fit for study participation
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH INTRAVENTRICULAR ADMINISTRATION OF HER2-CAR T CELLS: Participant has a released cryopreserved HER2-CAR T cell product
* ADDITIONAL ELIGIBILITY TO START CYCLE 1: Participant must have at least 1 metastatic brain lesion (measurable disease per RANO-Brain Metastases [BM] is not required-i.e., participant does not need to have at least 1 metastatic lesion >= 1 cm in longest dimension) that is new or increasing in size, or CSF cytology and/or radiographic findings consistent with leptomeningeal metastases
* ADDITIONAL ELIGIBILITY TO START CYCLE 1: Participants whose brain metastases have been treated with whole brain radiation (WBRT) or stereotactic radiosurgery (SRS): previously radiated metastases must have >= 20% increase in longest diameter that is also >= 5 mm absolute increase from prior brain MRI or histopathologically proven recurrent tumor. Otherwise, new or not previously radiated lesions must be present

  * Note: Participants who have undergone local therapy (surgical resection or biopsy, or SRS), must have recovered from all acute side effects before starting treatment with HER2-CAR T cells
* ADDITIONAL ELIGIBILITY TO START CYCLE 1: If a participant with brain metastases does not meet the above criteria, but there is still concern by the study team that changes in an enhancing brain lesion seen on brain MRI could be due to tumor progression, then the participant can undergo resection or biopsy of the lesion(s) to distinguish between tumor progression versus radiation necrosis. If there is histopathological evidence of tumor progression, then the participant can proceed with study treatment
* ADDITIONAL ELIGIBILITY TO START CYCLE 1: Research participant does not have uncontrolled seizure following surgery prior to starting the first CAR T cell dose
* ADDITIONAL ELIGIBILITY TO START CYCLE 1: Participants must have recovered from toxicity (=< grade 1) of prior therapy (excluding alopecia and peripheral neuropathy)
* ADDITIONAL ELIGIBILITY TO START CYCLE 1: Wash-out requirements (standard or investigational). The required waiting period between the last dose of the most recent chemotherapy agent(s) and first dose of HER2-CAR T cells is:

  * Four weeks for a cytotoxic chemotherapy, except for capecitabine, which will only require a 1 week waiting period from the last dose (on a dosing schedule of bid x 14 days, then off x 7 days);
  * At least 6 weeks must have passed since the completion of a nitrosourea-containing chemotherapy regimen;
  * At least four half-lives for a targeted agent

Exclusion Criteria:

* EXCLUSION CRITERIA FOR STUDY SCREENING: Research participant requires supplemental oxygen to keep saturation greater than 95% and the situation is not expected to resolve within 2 weeks
* EXCLUSION CRITERIA FOR STUDY SCREENING: Research participants with a known history of congestive heart failure (CHF) or cardiac symptoms consistent with NYHA classification III-IV within 6 months prior to day 1 of protocol treatment, cardiomyopathy, myocarditis, myocardial infarction (MI), exposure to cardiotoxic medications or with clinical history suggestive of the above must have an EKG and echocardiogram (ECHO) performed within 42 days prior to registration and as clinically indicated while on treatment.

  * Research participants with new symptoms of CHF, cardiomyopathy, myocarditis, MI, or exposure to cardiotoxic medications must have a cardiac consultation, creatinine phosphokinase (CPK), and troponin testing at pre study and as clinically indicated
* EXCLUSION CRITERIA FOR STUDY SCREENING: Research participant requires dialysis
* EXCLUSION CRITERIA FOR STUDY SCREENING: Research participant has uncontrolled seizure activity and/or clinically evident progressive encephalopathy
* EXCLUSION CRITERIA FOR STUDY SCREENING: Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase 1 study. A legal guardian may substitute for the research participant
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant is unwilling to stop treatment with chemotherapy or endocrine therapy during the first 3 cycles of the HER2-CAR T cell study
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant has a coagulopathy or bleeding disorder or cannot safely discontinue anticoagulation prior to placement of a Rickham reservoir
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant has a chronic or active viral infection of the CNS
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant has any uncontrolled illness, including ongoing or active infection; participant has known active hepatitis B or C infection; participants with any signs or symptoms of active infection, positive blood cultures or radiological evidence of infections
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant is human immunodeficiency virus (HIV) seropositive based on testing performed within 4 weeks of screening
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant has an autoimmune disease
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant has another active malignancy
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participants with lung metastases (exception may be allowed per principal investigator [PI] discretion for participants that are not symptomatic from their lung metastases)
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant is unable to undergo a brain MRI
* EXCLUSION CRITERIA FOR STUDY SCREENING: Participant is breast feeding. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with HER2-CAR T cells, breastfeeding should be discontinued if the mother wants to participate in this study
* EXCLUSION CRITERIA FOR STUDY SCREENING: Patient has a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the safety monitoring requirements and completion of treatment according to this protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | 21 days post T cell infusion
  Rate and associated 90% Clopper and Pearson binomial confidence limits (90% CI) will be estimated for participants' experiencing DLTs at the recommended phase 2 dose schedule.
Number of participants with treatment related adverse events | Up to 15 years
  Will be as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Tables will be created to summarize all toxicities and side effects by dose, time post treatment, organ, severity and arm.

SECONDARY OUTCOMES:
HER2-CAR T cells cerebrospinal fluid (CSF) and peripheral blood | Measured over time from baseline through 1 year, the number of measurements is determined by whether or not the participant has progressed (progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
Endogenous B cells in CSF and peripheral blood | Measured over time from baseline through 1 year, the number of measurements is determined by whether or not the participant has progressed (progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
T cells in CSF and peripheral blood | Progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
Myeloid cells in CSF and peripheral blood | Measured over time from baseline through 1 year, the number of measurements is determined by whether or not the participant has progressed (progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
Host immune subsets (e.g. T cell inhibitory/exhaustion markers, activation markers, and effector memory T cells) in CSF and peripheral blood | Measured over time from baseline through 1 year, the number of measurements is determined by whether or not the participant has progressed (progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
Cytokine levels in CSF | Measured over time from baseline through 1 year, the number of measurements is determined by whether or not the participant has progressed (progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
Cytokine levels in peripheral blood | Measured over time from baseline through 1 year, the number of measurements is determined by whether or not the participant has progressed (progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
Circulating tumor cells in the CSF | Measured over time from baseline through 1 year, the number of measurements is determined by whether or not the participant has progressed (progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Statistical and graphical methods will be used to describe the data.
Disease response in central nervous system (CNS) | Progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Will be evaluated by Response Assessment in Neuro-Oncology (RANO) criteria. Rates and 90% Clopper and Pearson Binomial Confidence limits will be calculated.
Systemic disease response | Progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Rates and 90% Clopper and Pearson Binomial Confidence limits will be calculated.
Median CNS progression-free survival | Progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)
  Kaplan Meier methods will be used.
Median overall survival | From time of surgery up to 15 years
  Kaplan Meier methods will be used.
HER2-CAR T cells detected in the tumor micro-environment | From time of surgery up to 15 years
  Statistical and graphical methods will be used to describe the data.
Immune cell subsets in the tumor micro-environment | From time of surgery up to 15 years
  Statistical and graphical methods will be used to describe the data.
Cytokine levels in the tumor micro-environment | From time of surgery up to 15 years
  Statistical and graphical methods will be used to describe the data.
HER2 antigen expression levels | From time of surgery up to 15 years
  Statistical and graphical methods will be used to describe the data.
Biomathematical modeling of tumor growth: perfusion and growth parameters based on serial brain magnetic resonance imaging | Progressed: baseline, 1, 3, 6, and 12 months, not progressed: baseline, 1, 3, 6, 8,10 and 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jana L Portnow, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States